CLINICAL TRIAL: NCT04604860
Title: EL-FIT (Exercise and Liver FITness): Validation of an Innovative Virtual Tool to Promote Physical Activity in Liver Transplant Candidates With Advanced Liver Disease
Brief Title: Use of EL-FIT App to Promote Physical Activity
Acronym: EL-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Association for the Study of Liver Diseases (AASLD) (Unknown); Pittsburgh Liver Research Center (Unknown)
Responsible Party: Principal Investigator, Andres Duarte-Rojo, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19020063
Record Dates: First submitted 2020-10-07; First posted 2020-10-27 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: End Stage Liver DIsease; Cirrhosis, Liver
MeSH Terms: conditions — End Stage Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EL-FIT (Experimental): Patients using the EL-FIT app
  Interventions: Behavioral: Fitness intervention

INTERVENTIONS:
Behavioral: Fitness intervention — Patients will follow exercise plans designed to promote physical activity (exercise and behavioral coaching).

SUMMARY:
Transplant-eligible patients with cirrhosis and ESLD, age 40-70, MELD >/= 10 referred to transplant physical therapy will be invited to participate. The investigators will exclude those who lack a smartphone or the understanding of its functionality, lack home wireless internet, or have recurrent/persistent overt hepatic encephalopathy. Following signing of informed consent, each participant will be given a Fitbit Charge 3 and have EL-FIT and Fitbit apps downloaded to their smartphone. After a brief session with a member of the research team explaining the basic components and functionality of EL-FIT and Fitbit, patients will be provided with general physical activity recommendations (as per our current standard of care) and asked to explore all features of EL-FIT and Fitbit apps, up until their 12-week follow-up visit. Phone calls to incentivize physical activity and exercise will be performed by members of the research team.

DETAILED DESCRIPTION:
The study consists of two visits, baseline and 12-week follow-up, with at least one follow-up phone call on a weekly basis. Visit one is expected to last for 30 minutes and visit 2 for 60 minutes, whereas each phone call should take no more than 15 minutes. Twice during the study period, the investigators will draw serum and plasma samples for future translational research. Daily, the physical trainer will review collected data on EL-FIT research database and Fitabase. Each participant will have an exit interview by the end of week 12 with the trainer and a member of the research team to talk about their impressions of using EL-FIT and Fitbit, through a structured questionnaire assessing about how user friendly it was to use the EL-FIT app. Finally, trainers will be asked to compare the type of prescription that they provided to patients as part of the standard of care (based on liver frailty index or 6-minute walk test), to compare it with the allocation provided by EL-FIT stratification algorithm.

To learn about how to improve EL-FIT the investigators will ask patients and their caregivers open-ended questions as part of their exit interview. This will allow us to identify barriers precluding them from keeping up with physical trainer recommendations, and what would they like to include to enhance motivation as part of a physical activity program. A member of the research team will act as a facilitator during this session.

ELIGIBILITY:
Inclusion Criteria:

* cirrhosis and ESLD
* transplant eligible
* MELD >/=10
* referred to transplant physical therapist

Exclusion Criteria:

* those who lack a smartphone or the understanding of its functionality
* lack home wireless internet
* have recurrent/persistent overt hepatic encephalopathy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Change in liver frailty index (LFI) score | 12 weeks
  Change in liver frailty index from baseline to the end of the study
Change in six minute walk test (6MWT) | 12 weeks
  Change in six minute walk test from baseline to the end of the study

SECONDARY OUTCOMES:
Change in daily average steps | 12 weeks
  Comparison of average daily steps from baseline until the end of study
Usability of EL-FIT app | 12 weeks
  How patient interacts with each of the features of EL-FIT app based on responses to questionairre

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No